CLINICAL TRIAL: NCT06219018
Title: The Effect of Medical Grade Honey (L-Mesitran) for Cervical Intraepithelial Neoplasia-II
Brief Title: Effect of Honey For CIN II
Acronym: HoneyForCINII
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL86044.096.23
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Cervical Intraepithelial Neoplasia-II; High Risk Human Papillomavirus
Keywords: Honey CINII

STUDY DESIGN:
Intervention Model Description: In this pilot study, we will include 60 patients with newly diagnosed CIN II. Patients will be counseled according to standard guidelines between a LLETZ, imiquimod or expectant management. Patients choosing for expectant management will be asked to participate in the study and will be treated with medical grade honey. Patients choosing for expectant management but not participating in the study and thus not using medicinal honey will be asked for the control arm. Follow-up assessment takes place in accordance with the national guideline (first check-up is after 6 months). In addition, swabs for vaginal microbiota analysis will be taken at 0 and 6 months. Immunohistochemical stainings for the local immune infiltrate will be performed on biopsies taken during regular colposcopy at t=0. This exploratory study aims to investigate the potential effect of honey and provides insight into its mechanisms of action.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Medical grade honey formulation (MGH) (L-Mesitran®) for CIN II (Experimental): Daily application of 5 grams (with applicator) for 3 months. Then weekly application (5 grams with applicator) for 3 months.
  Interventions: Drug: Medical grade honey formulation (MGH) (L-Mesitran®)

INTERVENTIONS:
Drug: Medical grade honey formulation (MGH) (L-Mesitran®) — Daily application of 5 grams (with applicator) for the first 3 months, followed by weekly application of 5 grams for the following 3 months.

SUMMARY:
The following hypothesis is tested: Medical grade honey in CIN II causes a higher clearance of the hr-HPV virus and an increase in the normalization of CIN II lesions compared to expectant management.

DETAILED DESCRIPTION:
In this pilot study, we will include 60 patients with newly diagnosed CIN II. Patients will be counseled according to standard guidelines between a LLETZ, imiquimod or expectant management. Patients choosing for expectant management will be asked to participate in the study and will be treated with medical grade honey. Patients choosing for expectant management but not participating in the study and thus not using medicinal honey will be asked for the control arm. Follow-up assessment takes place in accordance with the national guideline (first check-up is after 6 months). In addition, swabs for vaginal microbiota analysis will be taken at 0 and 6 months. Immunohistochemical stainings for the local immune infiltrate will be performed on biopsies taken during regular colposcopy at t=0. This exploratory study aims to investigate if there is a potential effect of honey and provides insight into its mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-40 years
* Primary CIN II confirmed histologically in the biopsy on colposcopic examination
* Sufficient mastery of the Dutch language

Exclusion Criteria:

* Simultaneous abnormality in columnar epithelial cells (AIS).
* Hr-HPV negative cytology
* Immunosuppressant use/Autoimmune disease (HIV, CVID)
* History of cervical carcinoma or previous treatment for CIN (LLETZ or imiquimod)
* Pregnancy or the intention to become pregnant during the study period
* Legal incompetence
* Known allergies to honey

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Clearance of hr-HPV | 6 months
  The following hypothesis is tested: Medical grade honey in CIN II causes a higher clearance of the hr-HPV virus

SECONDARY OUTCOMES:
Regression of CIN II | 12-24 months
  Defined as a regression to Pap 1
Clearance of hr-HPV and normalization of cytology (KOPAC) | 12-24 months
  Normalization of cytology (KOPAC) (depending on NVOG/RIVM flowchart).
Characteristics of the vaginal microbiome | 0-6 months
  Species specific and diversity analysis, changes due to honey and relationship with the other outcomes measures
Cervical immune status | 0 months
  Immunohistochemical stains on colposcopy biopsies for T and Myeloid cells
Human vaginal gene expression profiles | 0 and 6 months
  RNA quantity and quality of 20 patients
Quality of life, side-effects and compliance with medical grade honey | 0, 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Zuyderland MC, Heerlen, Limburg
  - Maastricht University Medical Centre+, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be shared.
Supporting Information: Study Protocol
Time Frame: Data will be available after publication of results.
Access Criteria: The data sharing plan includes that data (deidentified participant data) is available upon reasonable request from the corresponding author. This data could be used for further research or a meta-analysis on the use of medical grade honey for CIN II lesions. Data will be available after publication of results. Data can be available from the corresponding author J.N.M.M. Prop (https://orcid.org/0009-0009-8506-5797).'

REFERENCES:
- [Derived] Prop J, De Vos van Steenwijk P, Lardenoije CMJG, Cremers NAJ, Morre SA, Mongula J. Effect of medical-grade honey (L-Mesitran) for cervical intraepithelial neoplasia II: protocol for a multicentre cohort pilot study (HONEY FOR CIN II study). BMJ Open. 2025 Jul 24;15(7):e104585. doi: 10.1136/bmjopen-2025-104585. PMID 40707147